CLINICAL TRIAL: NCT01050569
Title: Innovative Interventions for Smoking Cessation: Comparison of Very Low Nicotine Content Cigarettes Plus Nicotine Patch; Very Low Nicotine Content Cigarettes Alone or Nicotine Patch Alone
Brief Title: Innovative Interventions for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0409M63686; 1R01DA025598 (NIH)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation; Nicotine Free Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VLNC Cigarette (Active Comparator): Very Low Nicotine Content Cigarette. Dosage: 0.05 mg to 0.09 mg nicotine yield cigarette; Frequency: Daily; Duration: 6 weeks.
  Interventions: Other: VLNC Cigarette
- Nicotine Patch (Active Comparator): 21 mg nicotine patch. Dosage: 21 mg; Frequency: Daily; Duration: 6 weeks.
  Interventions: Drug: Nicotine Patch
- VLNC Cigarette plus Nicotine Patch (Experimental): Very Low Nicotine Content Cigarette plus 21 mg Nicotine Patch. Patch Dosage: 21 mg; Cigarette Dosasge: 0.05 to 0.09 mg nicotine yield; Frequency: Daily; Duration: 6 weeks
  Interventions: Other: VLNC Cigarette Plus Nicotine Patch

INTERVENTIONS:
Drug: Nicotine Patch — 21 mg
  Other Names: Nicoderm CQ
  Arms: Nicotine Patch
Other: VLNC Cigarette — Cigarette where the tobacco contains <0.1 mg of nicotine yield.
  Other Names: Quest 3; Xodus
  Arms: VLNC Cigarette
Other: VLNC Cigarette Plus Nicotine Patch — 21 mg nicotine patch plus use of cigarette with tobacco containing <0.1 mg nicotine yield.
  Other Names: Nicoderm CQ; Quest 3; Xodus
  Arms: VLNC Cigarette plus Nicotine Patch

SUMMARY:
The purpose of this study is to evaluate the effect of a combination of the 21 mg nicotine patch and very low nicotine content (VLNC) cigarettes compared to 21 mg nicotine patch only and very low nicotine content cigarette only on abstinence, time to relapse and toxicant levels. The study will determine if adding nicotine replacement medication to the very low content cigarettes (VLNC) will augment treatment compared to nicotine patch only or to very low nicotine content cigarettes only.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of a combination of the 21 mg nicotine patch and very low nicotine content cigarette (VLNC) compared to the VLNC cigarette alone or 21 mg nicotine patch alone on abstinence, time to relapse and toxicant levels.

The following primary hypothesis will be tested:

Abstinence rates will be highest and the time to relapse will be the longest in the VLNC cigarettes plus nicotine patch condition compared to nicotine patch or VLNC cigarettes alone.

Other hypotheses include:

1. Greater positive subjective responses to cigarettes will be observed with VLNC cigarettes plus patch vs. VLNC cigarette;
2. Less drop-outs will be observed in the VLNC plus patch vs the other two conditions; and
3. Less compensatory smoking will be observed in the VLNC plus patch condition compared to VLNC cigarette alone condition.

Cigarette smokers will be randomized to:

1. VLNC cigarettes (which provide sensory behavioral aspects of smoking but with limited nicotine) plus nicotine patch for 6 weeks;
2. Nicotine patch for 6 weeks; or
3. VLNC cigarettes alone.

Outcome measures will include cessation assessed at the end of treatment as the primary endpoint and at 36 weeks post-treatment, time to lapse and relapse to usual brand cigarettes, and biomarkers of toxicant exposure. Predictors of abstinence and treatment response for each of the treatment conditions will be explored.

ELIGIBILITY:
Inclusion Criteria:

* a) Smoking at least 10 cigarettes daily for the past year;
* b) In good physical health;
* c) No contraindications for medicinal nicotine; and
* d) Stable, good mental health.

Exclusion Criteria:

* a) Subjects must not be using other tobacco or nicotine products.
* b) Female subjects cannot be pregnant or nursing and must be using appropriate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Duluth, Minnesota
  - University of MN's Tobacco Use Research Center, Minneapolis, Minnesota

REFERENCES:
- [Result] Hatsukami DK, Hertsgaard LA, Vogel RI, Jensen JA, Murphy SE, Hecht SS, Carmella SG, al'Absi M, Joseph AM, Allen SS. Reduced nicotine content cigarettes and nicotine patch. Cancer Epidemiol Biomarkers Prev. 2013 Jun;22(6):1015-24. doi: 10.1158/1055-9965.EPI-12-1439. Epub 2013 Apr 19. PMID 23603206
- [Derived] Dermody SS, Donny EC, Hertsgaard LA, Hatsukami DK. Greater reductions in nicotine exposure while smoking very low nicotine content cigarettes predict smoking cessation. Tob Control. 2015 Nov;24(6):536-9. doi: 10.1136/tobaccocontrol-2014-051797. Epub 2014 Sep 5. PMID 25192771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Oct 2008 to September 2011 Location was at the University of Minnesota Twin Cities and Duluth, Minnesota
Pre-assignment Details: After signing consent and before randomization to groups, 44 were lost to follow-up, 17 were ineligible, 10 were no longer interested, 10 were family members of enrollees.
Groups:
- VLNC Cigarette: Very Low Nicotine Content Cigarette: Cigarette where the tobacco contains <0.1 mg of nicotine yield. Participants were asked to smoke experimental cigarettes in an ad lib basis. Product was used for 6 weeks.
- VLNC Cigarette Plus Nicotine Patch: Very Low Content Cigarette Plus Nicotine Patch: 21 mg nicotine patch plus use of cigarette with tobacco containing <0.1 mg nicotine yield. Nicotine patch was administered on a daily basis. Participants were asked to use experimental cigarettes on an ad lib basis. Products were used for 6 weeks.
- Nicotine Patch: Nicotine Patch: 21 mg. Nicotine patch was administered on a daily basis for a period of 6 weeks.
Period: Overall Study
Arm/Group | VLNC Cigarette | VLNC Cigarette Plus Nicotine Patch | Nicotine Patch
Started | 79 | 76 | 80
Completed | 41 | 52 | 47
Not Completed | 38 | 24 | 33
Not completed — Lost to Follow-up | 20 | 14 | 16
Not completed — Withdrawal by Subject | 9 | 3 | 11
Not completed — Lack of Efficacy | 5 | 4 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- VLNC Cigarette: Very Low Nicotine Content Cigarettes : Cigarette where the tobacco contains <0.1 mg of nicotine yield.
- Nicotine Patch: 21 mg nicotine patch
- Total: Total of all reporting groups
Arm/Group | VLNC Cigarette | VLNC Cigarette Plus Nicotine Patch | Nicotine Patch | Total
Number analyzed (Participants) | 79 | 76 | 80 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 74 | 76 | 225
  >=65 years | 4 | 2 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.2) | 47.0 (11.9) | 47.3 (11.0) | 47.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 46 | 136
  Male | 32 | 33 | 34 | 99
Region of Enrollment [Number; unit: participants]
  United States | 79 | 76 | 80 | 235

OUTCOME MEASURES:

1. Primary Outcome: End of Treatment Abstinence Rate
Description: Cotinine and carbon monoxide (CO) verified point prevalence abstinence
Time Frame: 12 week
Measure: Number; unit: participants
Groups:
- VLNC Cigarette: VLNC Cigarettes: Cigarette where the tobacco contains <0.1 mg nicotine yield.
- VLNC Cigarette Plus Nicotine Patch: Very Low Nicotine Cigarette Plus Nicotine Patch: 21 mg nicotine patch plus use of cigarette with tobacco containing <0.1 mg nicotine yield.
Arm/Group | VLNC Cigarette | VLNC Cigarette Plus Nicotine Patch | Nicotine Patch
Number analyzed (Participants) | 79 | 76 | 80
participants | 19 | 18 | 19

2. Primary Outcome: End of Follow-up Abstinence Rates
Description: CO- and cotinine-verified point prevalence abstinence
Time Frame: 36 weeks
Measure: Number; unit: participants
Groups:
- VLNC Cigarette: Very Low Nicotine Content Cigarettes: Cigarette where the tobacco contains <0.1 mg of nicotine yield.
- VLNC Cigarette Plus Nicotine Patch: Very Low Nicotine Content Cigarette Plus Nicotine Patch: 21 mg nicotine patch plus use of cigarette with tobacco containing <0.1 mg nicotine yield.
Arm/Group | VLNC Cigarette | VLNC Cigarette Plus Nicotine Patch | Nicotine Patch
Number analyzed (Participants) | 79 | 76 | 80
participants | 14 | 15 | 15

3. Secondary Outcome: Exposure to Tobacco Toxicants
Time Frame: 6 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mg creatinine
Groups:
- VLNC Cigarette Plus Nicotine Patch: Very Low Nicotine Content Cigarette Plus Nicotine Patch : 21 mg nicotine patch plus use of cigarette with tobacco containing <0.1 mg nicotine yield.
Arm/Group | VLNC Cigarette | VLNC Cigarette Plus Nicotine Patch | Nicotine Patch
Number analyzed (Participants) | 52 | 55 | 59
pmol/mg creatinine
  Urinary 4-(methylnitrosamino)-1-(3-pyridyl)-1-buta | 0.40 [0.29 to 0.55] | 0.26 [0.19 to 0.36] | 0.25 [0.18 to 0.34]
  Total Nicotine Exposure (TNE) | 6.89 [4.26 to 11.02] | 27.39 [17.29 to 43.38] | 23.10 [14.59 to 36.60]
  Cotinine | 2.03 [1.20 to 3.45] | 7.65 [4.59 to 12.76] | 5.50 [3.31 to 9.13]

4. Secondary Outcome: Time to Lapse or Relapse to Tobacco Use
Time Frame: 26 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- VLNC Plus Nicotine Patch: Very Low Nicotine Content Cigarette Plus Nicotine Patch: 21 mg nicotine patch plus use of cigarette with tobacco containing <0.1 mg nicotine yield.
Arm/Group | VLNC Cigarette | VLNC Plus Nicotine Patch | Nicotine Patch
Number analyzed (Participants) | 78 | 76 | 80
weeks | 2.6 [1.7 to 5.9] | 7.1 [6.7 to 7.7] | 2.1 [1.6 to 3.9]

ADVERSE EVENTS:
Arm/Group | VLNC Cigarette | VLNC Cigarette Plus Nicotine Patch | Nicotine Patch
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/76 | 0/80
Other Adverse Events (participants affected / at risk) | 60/79 | 56/76 | 54/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLNC Cigarette (N=79) | VLNC Cigarette Plus Nicotine Patch (N=76) | Nicotine Patch (N=80)
Dry Mouth (General disorders) | 26 (42) | 25 (55) | 14 (26)
Headaches (General disorders) | 21 (26) | 21 (25) | 19 (29)
Tachycardia (Cardiac disorders) | 3 (3) | 7 (7) | 7 (7)
Dizziness (Ear and labyrinth disorders) | 8 (9) | 13 (13) | 13 (13)
Lightheadedness (General disorders) | 11 (13) | 10 (12) | 10 (12)
Nausea (Gastrointestinal disorders) | 9 (14) | 14 (18) | 14 (18)
Stomach Ache (Gastrointestinal disorders) | 4 (6) | 5 (5) | 9 (13)
Constipation (Gastrointestinal disorders) | 11 (15) | 10 (20) | 7 (14)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 7 (8) | 5 (6)
Shakiness (General disorders) | 6 (6) | 6 (7) | 4 (4)
Belching (General disorders) | 5 (7) | 2 (2) | 8 (10)
Sore Throat (General disorders) | 14 (26) | 11 (14) | 5 (9)
Anxiety (Psychiatric disorders) | 13 (15) | 6 (8) | 13 (15)
Sleep Disturbance (General disorders) | 19 (28) | 38 (100) | 43 (90)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (29) | 15 (20)

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No